CLINICAL TRIAL: NCT05490823
Title: Validation of a Smartphone App for Anemia Screening Among General Population: A Clinical Trial
Brief Title: Validation of a Smartphone App for Anemia Screening Among General Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AnemiaApp-2021
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Anemia
Keywords: Smartphone app; Artificial intelligence; Public health
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients for app-based anemia screening (Experimental): Device: A smartphone app for anemia screening This app can achieve automatic detection of anemia based on patient-sourced images of fingernails and conjunctivae.
  Interventions: Device: A smartphone app for anemia screening

INTERVENTIONS:
Device: A smartphone app for anemia screening — This app can achieve automatic detection of anemia based on patient-sourced images of fingernails and conjunctivae.

SUMMARY:
The current standard for anemia screening, complete blood count, presents invasiveness, infrastructure requirements and high costs, leading to serious underestimation of anemia prevalence and insufficient care for anemia patients. Here, the investigators established and validated an artificial intelligence system to achieve automatic detection of anemia based on patient-sourced images of fingernails and conjunctivae. This system has been integrated into a smartphone app to be further validated through hospital-based and population-based clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be aware of the contents and signed for the informed consent.

Exclusion Criteria:

* Patients who underwent ophthalmic or fingernail surgery in the past 30 days

Ages: 3 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of accurate, mistaken and missed detection of this smartphone app. | 27 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China